CLINICAL TRIAL: NCT03671603
Title: The Association of Iodixanol (Visipaque) to Renal Function and Cardiac and Cerebrovascular Events in STEMI Patients Undergoing Primary PCI: A Prospective, Multi-National, Multi-Center, Open-Label, Observational Study
Brief Title: Post-Marketing Safety Study in ST-Segment Elevation Myocardial Infarction (STEMI) Participants Undergoing Primary Percutaneous Coronary Intervention (PCI) Procedure With VISIPAQUE® as the Contrast Medium
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: VIS-16-07; VIS-16-07 (Other: GE HealthCare)
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Disease; ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction | interventions — iodixanol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Iodixanol: Participants will receive Iodixanol 270 mg I/ml or Iodixanol 320 mg I/ml injection as a part of routine clinical practice at the medical discretion of the physician.
  Interventions: Drug: Iodixanol

INTERVENTIONS:
Drug: Iodixanol — Iodixanol 270 mgI/ml or 320 mg I/ml injection will be administered as part of clinical practice according to the judgment of the site with regard to medical need.
  Other Names: VISIPAQUE®

SUMMARY:
The purpose of this study is to prospectively observe the incidence rate of acute kidney injury (AKI), major adverse renal and cardiovascular events (MARCE) in participants who were diagnosed with ST-segment elevation myocardial infarction (STEMI) and have completed primary percutaneous coronary intervention (PCI) procedure following an injection of iso-osmolar contrast medium iodixanol (Visipaque) during the in-hospital period and up to 30 days post-PCI follow-up period. The study will provide a better safety profile of Visipaque as the contrast medium in PCI procedure.

ELIGIBILITY:
Inclusion Criteria:

Participants may be included in the study if they meet all of the following criteria:

* The participant is over 18 years' old
* The participant with ST segment elevation myocardial infarction (STEMI) diagnosis has completed primary percutaneous coronary intervention (PCI) procedure and Visipaque was used as the contrast medium in the procedure
* The participant completed pre-procedural serum creatinine (SCr) test at the same hospital where PCI procedure was conducted, and the SCr test should be conducted with the same methodology before and after the procedure
* The participant has signed and dated the written informed consent form

Exclusion Criteria:

Participants must be excluded from participating in this study if they meet any of the following criteria:

* The participant has any contraindications to Visipaque (e.g., manifest thyrotoxicosis, history of serious hypersensitivity reaction to iodinated contrast media)
* The participant is pregnant or lactating
* The participant has been previously enrolled in this study
* The participant is currently under renal dialysis
* The participant presents with a terminal (life expectation <1 month), serious, or life-threatening disease, or any medical or psychiatric condition, or any condition where study participation may compromise the management of the participant
* The participant has other reasons that in the judgement of the investigator is unsuitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adult participants with STEMI diagnosis and have completed primary PCI procedure using Visipaque as contrast medium. The participants should complete pre-procedural SCr test at the same hospital where PCI procedure was conducted, and the SCr test should be conducted with the same methodology before and after the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 2755 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Assessment of the Incidence Rate of AKI in STEMI Participants Undergoing Primary PCI Using Visipaque | Within 48-72 hours post PCI
  AKI which is defined as a serum creatinine (SCr) increase of ≥ 0.3 mg/dL (≥ 26.4 umol/L) or increase to ≥150% (≥1.5-fold) from baseline values within 48-72 hours.

SECONDARY OUTCOMES:
Assessment of the Incidence Rate of MARCE in STEMI Participants Undergoing Primary PCI Using Visipaque Within 72 Hours Post-PCI | Within 72 hours post-PCI
  MARCE includes cardiac death, re-infarction, target lesion revascularization (TLR), stent thrombosis, unstable angina, stroke, transient ischemic attack (TIA), AKI, renal failure requiring dialysis.
Assessment of the Incidence Rate of Each Event of MARCE (except AKI) in STEMI Participants Undergoing Primary PCI Using Visipaque Within 72 Hours Post-PCI | Within 72 Hours post-PCI
  MARCE includes cardiac death, re-infarction, TLR, stent thrombosis, unstable angina, stroke, TIA, AKI, renal failure requiring dialysis.
Assessment of the Incidence Rate of MARCE (Except AKI) in STEMI Participants Undergoing Primary PCI Using Visipaque From 72 hours to 30 days Post-PCI | From 72 hours to 30 days post-PCI
  MARCE includes cardiac death, re-infarction,TLR, stent thrombosis, unstable angina, stroke, TIA, AKI, renal failure requiring dialysis.
Assessment of the Incidence Rate of Each Event of MARCE (except AKI) in STEMI Participants Undergoing Primary PCI Using Visipaque From 72 hours to 30 Days Post-PCI | From 72 hours to 30 Days post-PCI
  MARCE includes cardiac death, re-infarction, TLR, stent thrombosis, unstable angina, stroke, TIA, AKI, renal failure requiring dialysis.
All-Cause Mortality of STEMI Participants Within 30 days after primary PCI | From Baseline up to 30 days post-PCI

CONTACTS AND LOCATIONS:
Locations (36):
- China (35):
  - Kaifeng Central Hospital, Kaifeng, Contact:
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Dongguan Kanghua Hospital, Guangdong, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Shijiazhuang First Hospital Central Hospital Campus, Shijiazhuang, Hebei
  - Shijiazhuang First Hospital, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of CM, Zhengzhou, Henan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Wuhan Central Hospital, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - People's Hospital of Jiangsu Province, Nanjing, Jiangsu
  - China-Japan Friendship Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Ankang City Central Hospital, Ankang, Shaanxi
  - Linzi District People's Hospital, Linzi, Shandong
  - Shanxi Province Fenyang Hospital, Fenyang, Shanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Taiyuan Central Hospital, Taiyuan, Shanxi
  - Xi'an No.3 Hospital, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Ningbo First People's Hospital, Ningbo, Zhejiang
  - Shaoxing Hospital of Zhejiang University, Shaoxing, Zhejiang
  - Peking University First Hospital, Beijing
  - Wangjing Hospital of CACMS, Beijing
  - Shanghai Tongren Hospital, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai
  - Tianjin Chest Hospital, Tianjin
- Seoul National University Bundang Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No